CLINICAL TRIAL: NCT00359242
Title: Primary Prevention of Obesity Through Infancy Interventions
Brief Title: The SLeeping and Intake Methods Taught to Infants and Mothers Early in Life (SLIMTIME) Project
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Gerber Products Company (Industry)
Responsible Party: Principal Investigator, Ian M. Paul, MD, Professor of Pediatrics and Public Health Sciences Chief, Division of Academic General Pediatrics Vice Chair of Clinical Affairs, Department of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 22165EP; Grant Number: R56DK072996
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Weight Gain; Obesity
Keywords: Infant Sleep; Infant Diet; Infant Temperament; Rapid Infant weight gain; Infant Development; Parenting Competence; infant weight gain
MeSH Terms: conditions — Weight Gain; Obesity

ARMS (4):
- 1 (Experimental): Soothing and Calming instructions given at 2 weeks of life
  Interventions: Behavioral: Infant Sleeping and Soothing
- 2 (Experimental): Repeated food exposure instructions given between 4 and 6 months of life
  Interventions: Behavioral: Repeated Food Exposure
- 3 (Experimental): Receive both interventions: Soothing and Calming and Repeated food exposure
  Interventions: Behavioral: Infant Sleeping and Soothing; Behavioral: Repeated Food Exposure
- 4 (No Intervention): Group receiving neither of the interventions.

INTERVENTIONS:
Behavioral: Infant Sleeping and Soothing — Soothing and Calming instructions given to parents at a home visit when their infant is approximately 2 weeks old.
  Arms: 1; 3
Behavioral: Repeated Food Exposure — Instructions given to parents on introduction of solid foods and repeated exposure when the infant is approximately 4 to 6 months of age.
  Arms: 2; 3

SUMMARY:
Childhood obesity has reached epidemic proportions and its prevalence continues to rise, even among very young children. Because the current evidence base regarding potentially effective early intervention components to prevent obesity is so incomplete, it is logical to initiate obesity prevention intervention research during infancy, focusing on the two major components of the infant lifestyle, sleeping and feeding.

DETAILED DESCRIPTION:
Rationale: Childhood obesity has reached epidemic proportions and its prevalence continues to rise, even among very young children. A recent report from the National Health and Nutrition Examination Survey (NHANES) revealed that between 2003-2004, a staggering 26.2% of children aged 2 to 5 years were already overweight or at-risk for overweight. As such, in the summary of the "Conference on Preventing Childhood Obesity," it was remarked that researchers should particularly consider the youngest of children when planning obesity related interventions. Because the current evidence base regarding potentially effective early intervention components is so incomplete, it is logical to initiate obesity prevention intervention research during infancy, focusing on the two major components of the infant lifestyle, sleeping and feeding.

Key Objectives:

Aim 1: To evaluate the effect of simple procedures, taught to parents in the home environment by visiting nurses, that trains parents to calm their infants and increase their nocturnal sleep duration, thereby influencing sleep duration, nocturnal feeding frequency, and weight gain during infancy.

Aim 2: To evaluate a simple training procedure for parents, taught in the home environment by visiting nurses, that promotes infants' acceptance of nutritious, developmentally appropriate weaning foods.

Aim 3: To evaluate the delivery of these behavioral interventions to parents by community based home health nurses.

Aim 4: To examine the effect of a soothing intervention designed to increase sleep duration on overall maternal regulation of emotion, self-regulation of emotion, and weight gain.

Study Population: 160 newborns and mothers that demonstrate intent to breastfeed during the newborn nursery stay will be recruited during the maternity hospitalization. Approximately 25-50 physicians from the university affiliated pediatric and family practices.

ELIGIBILITY:
Inclusion Criteria:

* > 34 0/7 weeks gestational age
* Discharged from the newborn nursery or neonatal intensive care unit (NICU) without significant neonatal morbidity
* Singleton infant
* Nursery or NICU stay of 7 days or less
* Primiparous mother
* Maternity stay of 7 days or less
* Pediatric primary care provider from one of 3 University-affiliated pediatric practices or University-affiliated family medicine practices
* Feeding human milk (breast milk) during the maternity/newborn stay with intent to continue to breastfeed after discharge
* English speaking mother.

Exclusion Criteria:

* Newborn nursery, NICU, or maternity stay > 7 days
* Exclusive formula feeding in the nursery or NICU
* Multiparous mother
* Any metabolic condition that requires feedings at precise intervals
* Gestational age of 33 6/7 weeks or less
* Presence of a congenital anomaly or neonatal condition that significantly affects a newborn's feeding (e.g. cleft lip or cleft palate) or sleeping (hyperexplexia - exaggerated startle reflex)
* Non-singleton newborn

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2006-06; Primary Completion 2008-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Percent of infants sleeping 5 consecutive hours at night at 2 months of age | 2.5 years

SECONDARY OUTCOMES:
Duration breastfed | 2 years
Rate of weight gain | 2.5 years
Self-regulation of emotion | 3 years
Timing of introduction of solids | 3 years
Infant dietary variety | 3 years
Maternal feeding style | 3 years
Infant temperament | 3 years
Body Composition | 3 years
Lab evaluation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Leann Birch, PhD, Principal Investigator — Penn State University; Ian M Paul, MD, MSc, Study Director — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Paul IM, Savage JS, Anzman SL, Beiler JS, Marini ME, Stokes JL, Birch LL. Preventing obesity during infancy: a pilot study. Obesity (Silver Spring). 2011 Feb;19(2):353-61. doi: 10.1038/oby.2010.182. Epub 2010 Aug 19. PMID 20725058
- See also: Penn State Milton S. Hershey Children's Hospital Pediatric Clinical Research Office — http://www.hmc.psu.edu/pedsclinicalresearch/index.htm
- See also: Penn State University Center for Childhood Obesity Research — http://www.hhdev.psu.edu/ccor/